CLINICAL TRIAL: NCT04219774
Title: Neurocognitive Impairment Assessment in Symptomatic Carotid Occlusion Recanalized Endovascularly
Brief Title: NeuroCognition After Carotid Recanalization
Acronym: NIA-SCORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00110125
Record Dates: First submitted 2019-12-31; First posted 2020-01-07 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-03

CONDITIONS: Cognition Disorder; Stroke; Occlusion Carotid
MeSH Terms: conditions — Cognition Disorders; Stroke | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: 1:1 randomization, 1 non-randomized active comparator arm
Who Masked: Outcomes Assessor
Masking Description: Prospective randomized open blinded end-point (PROBE) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Endovascular arm (Experimental): Subjects meet all inclusion criteria and were randomized to intervention
  Interventions: Procedure: Endovascular intervention
- Medical arm (Active Comparator): Subjects meet all inclusion criteria and were randomized to best medical management
  Interventions: Drug: Aspirin and Clopidogrel (maximal medical Therapy)
- Non-Randomized Arm (Active Comparator): Subject meets all inclusion criteria EXCEPT abnormal CTP. Subjects are not randomized and are eligible for only best medical management
  Interventions: Drug: Aspirin and Clopidogrel (maximal medical Therapy)

INTERVENTIONS:
Procedure: Endovascular intervention — Endovascular angioplasty of the occluded carotid using balloon angioplasty and reconstruction with stents: coronary stents distally (Rebel, Boston Scientific; Vision, Abbott Vascular) and carotid stents proximal (Acculink and Xcat, Abbott Vascular) Patients will stay on their aspirin 325 mg and clopidogrel 75 mg
  Arms: Endovascular arm
Drug: Aspirin and Clopidogrel (maximal medical Therapy) — Best Medical Management: daily dual antiplatelet therapy (aspirin: 325 mg p.o. qd and Clopidogrel: 75 mg p.o. qd), optimization of systolic blood pressure (120 -140 mmHg), and smoking cessation.
  Arms: Medical arm; Non-Randomized Arm

SUMMARY:
Complete occlusion of the Internal carotid artery (ICA) by atherosclerotic disease (COICA) causes approximately 15%-25% of ischemic strokes in the carotid artery distribution. Patients treated with medical therapy have a 7%-10% risk of recurrent stroke per year for any stroke and a 5%-8% risk per year for ipsilateral ischemic stroke during the first 2 years after ICA occlusion. Internal carotid artery occlusion causes an estimated 61,000 first-ever strokes per year in the US an incidence more than twice the annual occurrence of ruptured intracranial aneurysms Additionally, 40% of subjects with COICA who present with transient ischemic attack (TIA) and 70% of COICA who present with stroke have cognitive decline with increased risk of vascular dementia and Alzheimer's' disease (AD) with time (2,3).

Symptomatic COICA subjects are at increased risk of developing cognitive impairment and progressive development of vascular dementia and AD with time. Our proposal leverages several compelling retrospective and prospective preliminary data from human to perform this exploratory trial with go/no-go criteria to proceed to a phase 3 based on the data generated

DETAILED DESCRIPTION:
Study Design:

Prospective randomized open blinded end-point (PROBE) study

This is a phase 2 randomized single-center open label clinical trial with randomization of 1:1 to either best medical management vs. best medical management and endovascular revascularization of COICA.

Screening, Enrolling, & Randomization:

All subjects who presents to our tertiary hospital with a diagnosis of COICA will undergo full evaluation including 1) documenting previous history of transient ischemic attack (TIA) and/or stroke; 2) cervical and brain CT angiography (CTA) to document complete occlusion; 3) CT perfusion (CTP) to assess for presence of penumbra evident by increased mean transient time (MTT) in the ipsilateral side of COICA; and 4) Montreal cognitive assessment (MoCA) score. If any subject is found to have complete occlusion of COICA, evident of abnormal/prolongation of MTT on CTP, previous history of TIA and or stroke, and MoCA <26 or abnormal response on another neuropsychological assessment preformed in the screening battery, then further evaluation is obtained including: MRI spectroscopy to assess for presence/absence of lactate in the ipsilateral watershed area (centrum semiovale), and size of ipsilateral hippocampus and amygdala, additional cognitive testing battery, and digital subtraction angiography (DSA) to document adequately the type of COICA the subject have (type A-D).

If a subject meets all inclusion criteria (complete occlusion, MoCA <26 and/or abnormal other neuropsychological test result, abnormal CTP) they will be randomized, after consent is obtained. If all inclusion criteria are met other than the CTP, they will be enrolled but not randomized. These subjects will only be eligible for best medical management- not surgical intervention.

If any subject does not have complete occlusion or abnormal MoCA >26 or other neuropsychological assessment, then the subject is excluded and no further testing needed (see exclusion criteria).

If the subject meets all inclusion criteria, then a baseline of complete neurological testing, full demographics, CTA or MRA, CTP, MoCA, additional neurological testing, MRI spectroscopy and DSA are obtained and subject is randomized 1:1 to either best medical management or best medical management + endovascular balloon angioplasty and stenting. Follow up clinic visits are arranged at 6 and 12 months. Repeat testing of MoCA and additional cognitive testing battery are done at these clinical follow-up visits (6 and 12 months). MRI of the brain and is done at 6 and 12 months. DSA is performed at 1 year follow-up for intervention subjects to assess brain bio-markers and revascularization respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Complete occlusion of cervical ICA on imaging studies (MRA or CTA) and confirmed with DSA
* History of TIA or stroke
* Increased MTT and/or time to peak (TTP) on CT perfusion as defined as T Max threshold of > 10cc > 4 seconds in the territory of the occluded carotid specifically in the MCA territory when compared to the opposite unaffected hemisphere (not required for observational cohort)
* All occlusion is due to atherosclerotic disease
* MoCA < 26 or abnormal result on another test in the battery (abnormal defined as 1.5 SD below age/ gender/ education matched norms).
* Baseline MoCA assessed by the neurosurgery team or neuropsychology team
* Failed best medical treatment (defined below)
* Class A and B on COICA Classification
* Study team able to gain consent from subject or legal adult representative (LAR)

Exclusion Criteria:

* Non-atherosclerotic occlusive disease that may have caused the occlusion, including moyamoya, dissection, trauma or other causes
* Tandem occlusion
* No evidence of penumbra on CT perfusion
* Severe co-morbid diseases: Chronic Kidney Disease (CKD) stages 4 or 5, end-stage renal disease, liver cirrhosis; Chronic Obstructive Pulmonary Disease (COPD) requiring home oxygen; terminal illness such as cancer; Parkinson disease or other neurodegenerative diseases; severe congestive heart failure; seizures; debilitating stroke, Modified Rankin Score (mRS) ≥ 3
* Short life expectancy due to cancer or other co-morbid diseases
* Class D on COICA classification
* Normal neuropsychological battery test results
* Subject unwilling to randomized to surgical procedure
* Pregnant or risk of becoming pregnant

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hasan, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of Iowa hospitals and Clinics, Iowa City, Iowa
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanaty M, Roa JA, Jabbour PM, Samaniego EA, Hasan DM. Recanalization of the Chronically Occluded Internal Carotid Artery: Review of the Literature. World Neurosurg X. 2019 Nov 21;5:100067. doi: 10.1016/j.wnsx.2019.100067. eCollection 2020 Jan. PMID 31872191
- [Background] Hudson JS, Zanaty M, Wadman V, Nakagawa D, Ishii D, Roa JA, Al Kasabz S, Limaye K, Rossen JD, Jabbour P, Adams HP Jr, Samaniego EA, Hasan DM. Bradycardia and Asystole in Patients Undergoing Symptomatic Chronically Occluded Internal Carotid Artery Recanalization. World Neurosurg. 2019 Nov;131:e211-e217. doi: 10.1016/j.wneu.2019.07.125. Epub 2019 Jul 23. PMID 31349074
- [Background] Limaye K, Zanaty M, Hudson J, Nakagawa D, Al Kasab S, Alvarez C, Dandapat S, Kung DK, Ortega-Gutierrez S, Jabbour P, Samaniego EA, Hasan D. The Safety and Efficacy of Continuous Tirofiban as a Monoantiplatelet Therapy in the Management of Ruptured Aneurysms Treated Using Stent-Assisted Coiling or Flow Diversion and Requiring Ventricular Drainage. Neurosurgery. 2019 Dec 1;85(6):E1037-E1042. doi: 10.1093/neuros/nyz226. PMID 31298301
- [Background] Zanaty M, Howard S, Roa JA, Alvarez CM, Kung DK, McCarthy DJ, Samaniego EA, Nakagawa D, Starke RM, Limaye K, Al Kasab S, Chalouhi N, Jabbour P, Torner J, Tranel D, Hasan D. Cognitive and cerebral hemodynamic effects of endovascular recanalization of chronically occluded cervical internal carotid artery: single-center study and review of the literature. J Neurosurg. 2019 Mar 29;132(4):1158-1166. doi: 10.3171/2019.1.JNS183337. Print 2020 Apr 1. PMID 30925474
- [Background] Zanaty M, Samaniego EA, Hasan DM. Letter to the Editor Regarding "Estimation and Recanalization of Chronic Occluded Internal Carotid Artery: Hybrid Operation by Carotid Endarterectomy and Endovascular Angioplasty". World Neurosurg. 2019 Jan;121:287. doi: 10.1016/j.wneu.2018.09.033. No abstract available. PMID 30557930
- [Background] Zanaty M, Samaniego EA, Teferi N, Kung DK, Nakagawa D, Hudson J, Ortega-Gutierrez S, Allan L, Jabbour P, Hasan DM. Hybrid Surgery for Internal Carotid Artery Revascularization. World Neurosurg. 2019 Jan;121:137-144. doi: 10.1016/j.wneu.2018.09.230. Epub 2018 Oct 9. PMID 30312821

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Arm: Participants without increased MTT or TPP on CTP may still be included in the unrandomized prospective observational arm.
Period: Overall Study
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Started | 12 | 13 | 6
6 Weeks Follow-up | 6 | 0 (The Medical arm did not have a 6-week follow-up visit.) | 6
6 Months Follow-up | 7 | 7 | 6
12 Months Follow-up | 6 | 4 | 6
Completed | 6 | 4 | 6
Not Completed | 6 | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm | Total
Number analyzed (Participants) | 12 | 13 | 6 | 31
Age, Continuous [Mean (Full Range); unit: years] | 65 [55 to 74] | 62 [47 to 86] | 60 [14 to 83] | 62 [41 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 0 | 5
  Male | 10 | 10 | 6 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 12 | 12 | 6 | 30
  Non-white | 0 | 1 | 0 | 1
  Latino and Hispanic | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 13 | 6 | 31
Medical History [Count of Participants; unit: Participants]
  Stroke | 9 | 10 | 4 | 23
  Current Hypertension | 9 | 9 | 3 | 21
  Transient Ischemic Attack | 6 | 5 | 2 | 13
  Carotid Artery Disease Surgery | 2 | 4 | 3 | 9
  Current COPD | 2 | 2 | 1 | 5
  Current Type 2 Diabetes Mellitus | 1 | 3 | 0 | 4
MoCA (Montreal Cognitive Assessment) Score [Count of Participants; unit: Participants] — The MoCA is a screening tool used to assess cognitive function. The possible score range is 0 to 30, with higher scores indicating better cognitive performance.
  Participants
    11-15 | 2 | 3 | 0 | 5
    16-20 | 2 | 1 | 1 | 4
    21-25 | 5 | 7 | 2 | 14
    26-29 | 3 | 2 | 3 | 8
Lesion Grade [Count of Participants; unit: Participants] — A: tapered occlusion of the ICA stump and patent lumen distally with collateral filling from branches of the ECA, posterior communicating artery (Pcom), and/or anterior communicating artery (ACA).
  B: nontapered ICA stump and patent lumen distally with collateral filling from branches of the ECA, Pcom, and/or ACA.
  C: no ICA stump and patent lumen distally with collateral filling, from branches of the ECA, Pcom, and/or ACA.
  D: no ICA stump and occluded lumen distally until the ICA bifurcation.
  Participants
    A | 5 | 4 | 1 | 10
    B | 2 | 3 | 0 | 5
    C | 5 | 6 | 5 | 16
    D | 0 | 0 | 0 | 0
Lesion Location [Count of Participants; unit: Participants]
  Left Internal Carotid Artery | 8 | 8 | 4 | 20
  Right Internal Carotid Artery | 3 | 3 | 2 | 8
  Bilateral Internal Carotid Artery | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Montreal Cognitive Assessment (MoCA) Score
Description: The MoCA is a screening tool used to assess cognitive function. The possible score range is 0 to 30, with higher scores indicating better cognitive performance.
Time Frame: Baseline, 6 months, 12 months
Population: Participants with data collected at both timepoints for each comparison.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 11 | 8 | 4
score on a scale
  Baseline to 6 months: number analyzed (Participants) | 9 | 8 | 4
  Baseline to 6 months | 0.56 (2.70) | 1.38 (2.83) | -0.75 (1.71)
  Baseline to 12 months: number analyzed (Participants) | 11 | 8 | 3
  Baseline to 12 months | 0.50 (2.20) | -0.80 (2.86) | -0.33 (1.15)

2. Primary Outcome: Change in Composite Cognitive Score
Description: This outcome reflects overall cognition. The composite z score is based on average z scores for the tests for each subject (sum of the z scores divided by the number of tests included) from a specifically designed battery of 14 cognitive tests: Montreal Cognitive Assessment (MoCA),Wide Range Achievement Test-5 (WRAT-5); Wechsler Adult Intelligence Scale - IV (WAIS-IV); WAIS-IV, Coding subtest; WAIS-IV, Matrix Reasoning subtest; Hopkins Verbal Learning Test; Benton Visual Retention Test (BVRT); Controlled Oral Word Association (COWA) Test; Boston Naming Test; Boston Diagnostic Aphasia Examination, Complex Ideational Material subtest; Trail-Making Test, part A and part B; Beck Depression Inventory-Fast Screen (BDI-FS); Iowa Scales of Personality Change (ISPC).
  A Z-score of 0 represents no change. Standard deviations above 0 represent better outcomes; standard deviations below 0 represent worse outcomes.
Time Frame: Baseline, 6 months, 12 months
Population: Participants with data collected at both timepoints for each comparison.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 9 | 8 | 3
z-score
  Baseline to 6 months: number analyzed (Participants) | 8 | 8 | 3
  Baseline to 6 months | 0.18 (0.63) | -0.005 (0.65) | 0.065 (0.88)
  Baseline to 12 months: number analyzed (Participants) | 8 | 7 | 2
  Baseline to 12 months | 0.36 (0.35) | 0.29 (0.76) | 0.26 (0.59)

3. Secondary Outcome: Number of Participants With Stroke Within 30 Days Post Procedure
Time Frame: Up to 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 12 | 13 | 6
Participants | 0 | 1 | 0

4. Secondary Outcome: Number of Participants With Intracranial Hemorrhage Within 72 Hours Post Procedure
Time Frame: Up to 72 hours post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 12 | 13 | 6
Participants | 1 | 0 | 0

5. Secondary Outcome: Number of Participant Deaths
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Observational: Participants without increased MTT or TPP on CTP may still be included in the unrandomized prospective observational arm.
Arm/Group | Endovascular Arm | Medical Arm | Observational
Number analyzed (Participants) | 12 | 13 | 6
Participants | 1 | 1 | 0

6. Other Pre Specified Outcome: Change in Mean Transit Time (MTT) on CT Perfusion
Description: MTT is defined as the average time, in seconds, that circulating blood cells needs to pass within a determinate volume of brain. It is assessed as part of the CT perfusion protocol.
Time Frame: Baseline, 12 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 10 | 9 | 3
seconds
  MTT - Left | 1.15 (0.51) | 1.46 (0.53) | 1.13 (0.1)
  MTT - Right: number analyzed (Participants) | 2 | 4 | 1
  MTT - Right | 0.60 (0.84) | 1.13 (0.95) | 1.14 (NA) — Only one participant analyzed

7. Other Pre Specified Outcome: Change in Size of Hippocampus
Description: The change in size of hippocampus in the ipsilateral side of COICA (t-test), at enrollment vs. 1 year.
Time Frame: Baseline, 6 months, 12 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 4 | 4 | 4
cm^3
  Hippocampus - Left (baseline to 6 months): number analyzed (Participants) | 4 | 1 | 4
  Hippocampus - Left (baseline to 6 months) | -67.54 (80.73) | 27.69 (0) | 49.08 (193.34)
  Hippocampus - Left (baseline to 12 months) | -69.00 (54.51) | -35.79 (78.42) | -77.62 (89.9)
  Hippocampus - Right (baseline to 6 months): number analyzed (Participants) | 4 | 1 | 4
  Hippocampus - Right (baseline to 6 months) | -54.92 (81.52) | 44.55 (0) | 43.05 (161.94)
  Hippocampus - Right (baseline to 12 months) | -102.30 (123.80) | -22.00 (45.24) | -83.44 (47.86)

8. Other Pre Specified Outcome: Change in Size of Amygdala
Description: The change in size of amygdala in the ipsilateral side of COICA (t-test), at enrollment vs. 1 year.
Time Frame: Baseline, 6 months, 12 months
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 4 | 4 | 4
cm^3
  Amydala - Left (baseline to 6 months): number analyzed (Participants) | 4 | 1 | 4
  Amydala - Left (baseline to 6 months) | -26.47 (60.02) | 33.89 (0) | 14.22 (19.74)
  Amydala - Left (baseline to 12 months) | -29.36 (52.95) | 2.85 (34.39) | -3.18 (5.68)
  Amydala - Right (baseline to 6 months): number analyzed (Participants) | 4 | 1 | 4
  Amydala - Right (baseline to 6 months) | -5.76 (22.27) | -0.64 (0) | 10.96 (24.65)
  Amydala - Right (baseline to 12 months) | -15.33 (6.61) | -2.26 (18.16) | -9.72 (15.06)

9. Other Pre Specified Outcome: Number of Participants With the Presence of Lactate on 1H-MRI Spectroscopy
Description: Presence of lactate determined by MRI spectroscopy in centrum semiovale in the ipsilateral side of chronic occlusion of the internal carotid artery (COICA).
Time Frame: Baseline, 6 months, 12 months
Population: Participants with data collected at each timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
Number analyzed (Participants) | 7 | 6 | 4
Participants
  Baseline | 1 | 3 | 0
  6 months: number analyzed (Participants) | 2 | 1 | 4
  6 months | 0 | 0 | 0
  12 months: number analyzed (Participants) | 2 | 2 | 4
  12 months | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Endovascular Arm | Medical Arm | Observational Arm
All-Cause Mortality (participants affected / at risk) | 1/12 | 1/13 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/12 | 6/13 | 3/6
Other Adverse Events (participants affected / at risk) | 10/12 | 8/13 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Arm (N=12) | Medical Arm (N=13) | Observational Arm (N=6)
Acute blood loss anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute systolic heart failure (Cardiac disorders) | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
EVD malfunction (Investigations) | 1 | 0 | 0
Expressive Aphasia (Nervous system disorders) | 1 | 0 | 0
Femoral Pseudoaneurysm (Blood and lymphatic system disorders) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Infarct (Cardiac disorders) | 1 | 0 | 0
Intraparenchymal hemorrhage (Cardiac disorders) | 1 | 0 | 0
Myelodysplastic Syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0
Perinephric hematoma (Blood and lymphatic system disorders) | 0 | 1 | 0
Posterior vitreous hemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0
Regressed neovascularization (Blood and lymphatic system disorders) | 0 | 1 | 0
Retroperitoneal hematoma (Blood and lymphatic system disorders) | 1 | 1 | 0
Stage 4 Urothelial cancer (Renal and urinary disorders) | 0 | 1 | 0
LICA (Cardiac disorders) | 1 | 0 | 0
Small bowel and Cecal AVM (Gastrointestinal disorders) | 1 | 0 | 0
Subacute Chronic Infarcts (Cardiac disorders) | 1 | 0 | 0
Subarachnoid hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0
Tonic Clonic Seizures (Nervous system disorders) | 1 | 0 | 0
Subclinical seizures (Nervous system disorders) | 1 | 0 | 0
Colon Re-section (Surgical and medical procedures) | 0 | 0 | 1
Lung mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mechanical Fall and Facial T (General disorders) | 0 | 0 | 1
Syncopal Fall (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Arm (N=12) | Medical Arm (N=13) | Observational Arm (N=6)
Acute blood loss anemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Altered mental status (Psychiatric disorders) | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Bloody Stool (Gastrointestinal disorders) | 0 | 1 | 0
Carpal Tunnel (General disorders) | 0 | 1 | 0
Cognitive Impairment (Psychiatric disorders) | 1 | 0 | 0
Decreased Mood (Psychiatric disorders) | 1 | 0 | 0
Diabetes Miletus (Endocrine disorders) | 1 | 0 | 0
Disorientation with Physical Effort (Investigations) | 2 | 0 | 0
Dissection of ECA (Cardiac disorders) | 1 | 0 | 0
Dysphasia (General disorders) | 1 | 0 | 0
Easy Bruising (General disorders) | 4 | 1 | 0
Excessive Bleeding (Blood and lymphatic system disorders) | 4 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Head trauma due to falls (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (General disorders) | 2 | 0 | 0
Hematuria (Blood and lymphatic system disorders) | 1 | 1 | 0
High Blood Pressure (Cardiac disorders) | 0 | 1 | 0
Hypotension (Cardiac disorders) | 4 | 0 | 0
Lactic acidosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Memory Impairment (Psychiatric disorders) | 1 | 1 | 0
Myocardial Injury (Cardiac disorders) | 1 | 0 | 0
Nose Bleeds (General disorders) | 1 | 0 | 0
Progressive Cognitive Impairment (Psychiatric disorders) | 0 | 1 | 0
Psychiatric Episode (Psychiatric disorders) | 1 | 0 | 0
Severe Anomia (Nervous system disorders) | 0 | 1 | 0
Transfusion Associated Circulatory Overload (Cardiac disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Vaginal bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Visual Field Deficit (Eye disorders) | 1 | 0 | 0
Wrist Hematoma (General disorders) | 1 | 0 | 0
Swelling in bilateral lower extremities (General disorders) | 1 | 0 | 0
Distal Interphalangeal Fract (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Essential Hypertension (Cardiac disorders) | 0 | 0 | 1
Shoulder Arthralgias (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Vision Changes (Eye disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The Observation Arm was not included in comparison. It is a non-equivalent group because patients included in the Arm if they were ineligible based on baseline measures and consent to randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04219774/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04219774/ICF_000.pdf